CLINICAL TRIAL: NCT02520271
Title: ODS is a Naturalistic, Open Label, Non-randomized Follow-up Study on Depression and Related Substance Use Disorders (SUD). Study Targets: Efficacy of Psychosocial Treatment, Pharmacogenetics, Inflammation Related Biomarkers
Brief Title: Ostrobothnia Depression Study (ODS). A Naturalistic Follow-up Study on Depression and Related Substance Use Disorders
Acronym: ODS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seinajoki Central Hospital (Other)
Collaborators: Tampere University (Other)
Responsible Party: Principal Investigator, Olli Kampman, Associate Professor, Seinajoki Central Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: EVO1114
Record Dates: First submitted 2015-06-27; First posted 2015-08-11 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Major Depression; Dual Diagnosis; Anxiety Disorders; Substance Related Disorders
Keywords: Mood Disorders; Motivational Interview; Behavioral Activation
MeSH Terms: conditions — Depressive Disorder, Major; Anxiety Disorders; Substance-Related Disorders; Mood Disorders | interventions — Cognitive Behavioral Therapy; Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Depression (Active Comparator): Behavioral activation only
  Interventions: Behavioral: Behavioral Activation
- Depression and SUD (Active Comparator): Motivational interview and Behavioral activation
  Interventions: Behavioral: Behavioral Activation; Behavioral: Motivational Interview

INTERVENTIONS:
Behavioral: Behavioral Activation — BA consists of at least 4 intervention sessions with a focused, active working style by the therapist. The therapy initiation includes a focused interview targeting at determining 1-2 main problems, on which the therapy will be focused. Specific therapeutic methods for BA include the use ABC analysis, targeting at hitting the negative consequences of current problematic behavior and motivating for change. Further, recognizing the obstacles for change (TRAP) is the next method to be used. The therapist encourages the client for active behavioral monitoring through assigned homework during the therapy process. The final step and method used is strengthening the gained change (ACTION).
  Other Names: Behavioral Activation Therapy; Cognitive Behavioral Therapy
Behavioral: Motivational Interview — Motivational interview (MI) is a therapeutic intervention that focuses on resolving client ambivalence towards changing problematic behavior. MI involves a client-centered approach that encourages the client to develop his or her own motivation. The therapeutic alliance in MI is predominantly a partnership, rather than an expert/client dynamic.
  MI has been studied primarily in addiction problems, but there are numerous reports of its efficacy in several chronic somatic conditions, and lifestyle problems.
  Other Names: Motivational Interviewing
  Arms: Depression and SUD

SUMMARY:
Ostrobothnia Depression Study (ODS) was conducted in the South Ostrobothnia hospital district of Finland during 2009-2014. ODS is a naturalistic, open label, non-randomized follow-up study on depression and related substance use disorders (SUD). The study focuses on several aspects concerning the relation of depression and SUDs, the efficacy of selected assessment and treatment protocols, characteristics and genetics of the participants and the use of related biomarkers in clinical practice. The misused substance in focus is alcohol. In this study, dual diagnosis (DD) is defined as the simultaneous presence of clinically diagnosed major depressive disorder (MDD) and alcohol use disorder (AUD). The study was approved by the local ethics committee. Written informed consent was collected from all participants.

DETAILED DESCRIPTION:
Participants The participants were recruited in five outpatient clinics and in one psychiatric hospital ward in the South Ostrobothnia hospital district (population 200,000) during 1.10.2009 - 31.10.2013. Patients referred to psychiatric secondary services because of depressive symptoms, anxiety, self destructiveness, insomnia and alcohol or other substance related problems were screened with Beck depression inventory (BDI, version 1A). Patients with BDI score ≥ 17 at the screening phase were recruited in the study. The patients with a likely or verified psychotic disorders (ICD-10, F2*.** diagnosis) or organic brain disease were excluded.

A total of 242 patients were included in the study. Fifty-three (21.9%) patients were hospitalised at baseline. The participants were aged 17-64 years (mean 38.8 years, SD 12.2). Among the recruited were 148 females (61.2%) and 94 males (38.8%). The Mini International Neuropsychiatric Interview 5.0 (MINI) was made at the baseline to 219 patients.

At baseline 203 (84%) patients were prescribed antidepressive medication, 81% of cases either SSRI or SNRI as primary antidepressant). Antipsychotic medication was prescribed to 66 (28%) patients.

At the time of recruitment the participants were divided in two groups based on the AUDIT -score. The patients with baseline AUDIT-score ≥ 11 were categorized as patients with comorbid AUD and therefore dual diagnosis (DD+). The patients with AUDIT ≤ 10 were categorized as (DD-).

The clinical psychiatric evaluation was performed by a psychiatrist or other trained professional using the Mini International Neuropsychiatric Interview 5.0 (MINI). The symptoms of MDD were assessed by the Montgomery-Åsberg Depression Rating Scale (MADRS).

The patients received medication if the need for medical treatment was assessed by the psychiatrist responsible of the treatment. The use of psychotropic medications was recorded. The choice of medication was left for the clinician in charge.

All participants were also evaluated by three-dimensional model to select the following treatment intervention. The model has been developed by Kampman and Lassila in South Ostrobothnia hospital district and described in more detail in Finnish Medical Journal. The model was developed based on the need to have tools to better assess the patients with DD in clinical setting. The model can be used for defining the patients' problem according to three treatment related factors (diagnosis, substance use problem, level of functioning). The model consists of three dichotomous assessments each leading to score of 0 or 1 points according to difficulty of the problem. The factors assessed are 1) psychiatric diagnosis (non-psychotic/psychotic; 0/1 points), 2) difficulty of SUD (moderate/difficult; 0/1 points) and 3) patients level of functioning according to Global Assessment of Functioning (GAF) -scale (good functioning/poor functioning; 0/1 points). The given points are then added together to form an overall score from 0 points (modest DD problem) to 3 points (most difficult DD problem).

Treatment interventions The treatment interventions included antidepressive medication (SSRI or other), Behavioral Activation therapy (BA) and FRAMES intervention, and Motivational interview (MI) In participants with AUDIT ≤ 10 (DD-) the intervention started with focus on depression (antidepressive medication and BA). In patients with AUDIT ≥ 11 (DD+) the intervention started with focus on AUD. If AUD was evaluated as moderate (duration less than 2 years, most of the days sober during the last month) the first treatment selected could be either FRAMES or MI. If AUD was assessed to be severe (duration more than 2 years, active use most of the days during last month, poly-substance use, GAF < 50) the intervention was supposed to start with MI. The intervention was implemented by the staff person responsible of the appointments of certain patient (a nurse or a psychologist) who had received training for the use of selected interventions. The duration of MI was set to approximately 3 (2-5) appointments. The minimum duration of BA was set to 4 appointments.

Follow-up The follow-up included appointments with clinical research nurse at 6, 12 and 24 months points. During these appointments the severity of and the recovery from depression was evaluated by MADRS, alcohol use was evaluated by AUDIT, the information on substance use relapses was collected, and the MINI-interview was repeated at 12 months point. Additionally, the following information was collected: 15D-quality of life scale, GAF-scale, laboratory tests (at 6 months: a blood count, electrolytes, creatinine, liver function), Body Mass Index, waist, smoking status.

ELIGIBILITY:
Inclusion Criteria:

Patients referred to psychiatric secondary services because of

1. Depressive symptoms
2. Anxiety
3. Self-destructiveness
4. Insomnia
5. Alcohol or other substance related problems, and had Beck depression inventory (BDI, version 1A) score at least 17 at the screening phase.

Exclusion Criteria:

* A likely or verified ICD-10 F2 category diagnosis (psychotic disorders).
* Organic brain disease

Ages: 17 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2009-10; Primary Completion 2013-10 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Change in severity of depressive symptoms from baseline at 6 weeks, 6 months, 12 months, and 24 months | baseline, 6 weeks, 6 months, 12 months, 24 months
  Measure: MADRS depression scale

SECONDARY OUTCOMES:
Change in quality of life from baseline at 6 weeks, 6 months, 12 months, and 24 months | baseline, 6 months, 12 months, 24 months
  Measure: 15D scale
Change in number of weekly consumed alcohol drinks from baseline at 6 weeks, 6 months, 12 months, and 24 months | baseline, 6 weeks, 6 months, 12 months, 24 months
Change in severity of alcohol use from baseline at 6 weeks, 6 months, 12 months, and 24 months | baseline, 6 weeks, 6 months, 12 months, 24 months
  Measure: AUDIT (Alcohol Use Disorders Identification Test)

CONTACTS AND LOCATIONS:
Overall Officials: Olli Kampman, MD, PhD, Study Director — Seinäjoki Hospital District, Department of Psychiatry and University of Tampere, School of Medicine
Locations (1):
- Seinäjoki Hospital District, Seinäjoki, South Ostrobothnia, Finland

REFERENCES:
- [Background] Miller WR, Rollnick S. Ten things that motivational interviewing is not. Behav Cogn Psychother. 2009 Mar;37(2):129-40. doi: 10.1017/S1352465809005128. PMID 19364414
- [Background] Kanter JW, Manos RC, Bowe WM, Baruch DE, Busch AM, Rusch LC. What is behavioral activation? A review of the empirical literature. Clin Psychol Rev. 2010 Aug;30(6):608-20. doi: 10.1016/j.cpr.2010.04.001. PMID 20677369
- [Background] Kampman O, Lassila A. Samanaikaisen mielenterveys- ja päihdeongelman hoitoon on kehitetty integroitu arviointimalli [TI: An Integrated Assessment Method for Dual Diagnosis]. Suom Lääkäril 2007:4447-4451.[SO: Finnish Medical Journal, Finnish]
- [Derived] Luoto KE, Lassila A, Leinonen E, Kampman O. Predictors of short-term response and the role of heavy alcohol use in treatment of depression. BMC Psychiatry. 2023 Nov 27;23(1):880. doi: 10.1186/s12888-023-05366-8. PMID 38012573
- [Derived] Archer M, Niemela O, Hamalainen M, Moilanen E, Leinonen E, Kampman O. The role of alcohol use and adiposity in serum levels of IL-1RA in depressed patients. BMC Psychiatry. 2022 Mar 2;22(1):158. doi: 10.1186/s12888-022-03784-8. PMID 35232419
- [Derived] Luoto KE, Lindholm LH, Koivukangas A, Lassila A, Sintonen H, Leinonen E, Kampman O. Impact of Comorbid Alcohol Use Disorder on Health-Related Quality of Life Among Patients With Depressive Symptoms. Front Psychiatry. 2021 Oct 8;12:688136. doi: 10.3389/fpsyt.2021.688136. eCollection 2021. PMID 34690824
- [Derived] Luoto KE, Lindholm LH, Paavonen V, Koivukangas A, Lassila A, Leinonen E, Kampman O. Behavioral activation versus treatment as usual in naturalistic sample of psychiatric patients with depressive symptoms: a benchmark controlled trial. BMC Psychiatry. 2018 Jul 27;18(1):238. doi: 10.1186/s12888-018-1820-x. PMID 30049272